CLINICAL TRIAL: NCT04859270
Title: The Holistic Health Care of Post-Cardiac Arrest Survivors: From Patient's Health to Family Resilience
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012242RINB
Record Dates: First submitted 2021-04-14; First posted 2021-04-26 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-02

CONDITIONS: Post-Cardiac Arrest Syndrome
Keywords: Post-cardiac arrest; Holistic care; Family resilience
MeSH Terms: conditions — Post-Cardiac Arrest Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Post-cardiac arrest mortality remains high and proper care after cardiopulmonary resuscitation is an important clinical challenge. This prospective observational cohort aims to (1) identify the factors that affect short-term and long-term survival in post-cardiac arrest survivors and (2) investigate the patients and their families' health-related quality of life and psychological well-being.

DETAILED DESCRIPTION:
For this cohort study, adult survivors (≧20 years) of sudden cardiac arrest for more than 5 minutes after cardiopulmonary resuscitation will be enrolled. Basic demographic information, clinical events throughout hospitalization, and laboratory examination results will be recorded. Patients will be assessed for their neurological outcome using Glasgow coma score (GCS) and cerebral performance categories (CPC) upon hospital discharge, 1, 3, 6, and 12 months after discharge.

Post-cardiac arrest care is clinically challenging and this study aims to evaluate not just the physical well-being but also the psychological well-being of these patients on the short-term and long-term survival. Patients and their families will be assessed on their health-related quality of life and psychological well-being upon hospital discharge using the following scales: Mayo-Portland Adaptability Inventory (MPAI-4), World Health Organization Quality of Life Scale (WHOQOL-BREF), Impact of Event Scale - Revised (IES-R), and Family Resilience Framework. They will also be followed for one year after discharge at 1, 3, 6, and 12 months.

Data will be analyzed using the SPSS and SAS package. Odds ratios and hazards ratios will be determined for the factors that affect survival after cardiac arrest. The findings will help clinicians provide timely support to the patients and their families to promote physical and psychological well-being, and integrate them back to society as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-traumatic cardiac arrest, who have successfully sustained return of spontaneous circulation for more than five minutes after resuscitation efforts.

Exclusion Criteria:

1. Under 20 years of age
2. Pregnant
3. Terminally ill cancer patients or cancer patients who are unwilling to receive treatment
4. When the ICU is over capacity and unable to provide intensive care.
5. The patient or family members refused to participate in this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary participants of the study are patients with out-of-hospital cardiac arrest and achieved return of spontaneous circulation after cardiopulmonary resuscitation. The number of primary participants is 200, and the interviewees are patients and their family members (400), a total of 600 participants.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Post-cardiac arrest survival | Up to 1 year after discharge
  Post-cardiac arrest survival after cardiopulmonary resuscitation
Neurological outcome - GCS | Up to 1 year after discharge
  Using the Glasgow Coma Scale (GCS) of the patients, with scores ranging from 3 to 15, and higher scores indicating a better outcome.
Neurological outcome - CPC | Up to 1 year after discharge
  Cerebral performance categories (CPC) of the patients, with categories 1 and 2 as favorable outcomes, and categories 3 to 5 as unfavorable outcomes
Functional outcome | Up to 1 year after discharge
  Self-reported assessment using the Mayo-Portland Adaptability Index (MPAI-4) for the patients. This is a 29-item scale with overall scores ranging from 0 to 111, and lower scores indicating a better outcome and greater community reintegration post-injury.
Life quality | Up to 1 year after discharge
  Self-reported assessment using the abbreviated World Health Organization Quality of Life questionnaire (WHOQOL-BREF) for the patients. This is a 26-item scale with overall transformed scores ranging from 0 to 100, and higher scores indicating a better quality of life.
Emotional stress | Up to 1 year after discharge
  Self-reported assessment using the Impact of Events Scale - Revised (IES-R) for the patients. This is a 22-item scale with scores ranging from 0 to 88, and higher scores indicating more subjective distress.
Family resilience | Up to 1 year after discharge
  Self-reported assessment using the Family Resilience Framework scale for the patients and their families. This is a 31-item scale with scores ranging from 0 to 155, and higher scores indicating a higher level of resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Shan Tsai, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No